CLINICAL TRIAL: NCT06046430
Title: Investigation of Laterality and Sensory Acuity Abilities of Frozen Shoulder Patients
Status: Completed | Type: Observational
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Principal Investigator, Harran University
Other Study IDs: 1
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Frozen Shoulder; Laterality Defects
MeSH Terms: conditions — Bursitis | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frozen Shoulder Group: The sample of the study will consist of patients who applied to Harran University Hospital and were diagnosed with frozen shoulder.
  Interventions: Other: Assessment
- Healthy Group: Healthy volunteers similar to the patient group in gender and age factors.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The same assessments will be made to participants in both groups.

SUMMARY:
The brain contains the body representation necessary for normal functioning, including goal-directed movements and behaviors. Body representation involves integrated sensory input and ideas about one's body. Both executed and imagined movements depend on the representation of the body in the cortical area. Laterilization is one of the motor imagery methods that requires activation of proprioceptive, somatosensory and premotor regions and enables the determination of pain-induced cortical changes. Another method to determine pain-related somatosensory changes is the two-point discrimination test.

It is suggested that laterization and sensory acuity responses may change due to long-term pain and stiffness experienced in people with frozen shoulders. Therefore, the aim of this study is to investigate the laterization and sensory acuity abilities of patients with frozen shoulder.

ELIGIBILITY:
Frozen Shoulder Group:

Inclusion Criteria:

Patients with shoulder pain of at least six months' duration secondary to tendinopathy and/or partial rotator cuff tear; Patients with ability to follow simple orders; iii) Patients with ability to sign to provide informed consent

Exclusion Criteria:

Normal passive ROM External ROM < 30 To have received treatment (physiotherapy, intra-articular injection, surgery) related to the existing complaint Pain < 3 according to the numbered pain assessment scale

Healthy group :

Inclusion criteria:

No actual shoulder pain or previous history of shoulder complaints including Frozen Shoulder.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample of the study will consist of patients who applied to Harran University Hospital and were diagnosed with frozen shoulder.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Right-Left Discrimination | Baseline
  Right-Left Discrimination will be assessed with Recognise™ application. It tests the patients' ability to quickly and accurately recognise an image of a body area as either left or right ('Left/Right Discrimination'). The test will be repeated three times and average values will be recorded.
Acuity | Baseline
  Two point discrimination is the ability to discern that two nearby objects touching the skin are truly two distinct points, not one.In clinical settings, two-point discrimination is a widely used technique for assessing tactile perception. It relies on the ability and/or willingness of the patient to subjectively report what they are feeling and should be completed with the patient's eyes closed. Aesthesiometer is the instrument used to determine two point discrimination values.

SECONDARY OUTCOMES:
Pain Intensity | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The higher scores indicate an higher level of pain.
Active Range of Motion (AROM) Assessment | Baseline
  The shoulder's AROM, including flexion, abduction, internal and external rotation will be measured described by the American Academy of Orthopaedic Surgeons (AAOS) using a universal goniometer. The process will be repeated three times in each direction, with the average value recorded.
Central sensitization | Baseline
  The Central Sensitisation Inventory (CSI) is a self-report outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS).
  The CSI consists of two parts.
  Part A includes 25 questions related to common CSS symptoms. Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression
Pain Catastrophizing | Baseline
  Pain catastrophizing is characterized by the tendency to magnify the threat value of a pain stimulus and to feel helpless in the presence of pain, as well as by a relative inability to prevent or inhibit pain-related thoughts in anticipation of, during, or following a painful event. As such, the Pain Catastrophizing Scale (PCS) was developed to help quantify an individual's pain experience, asking about how they feel and what they think about when they are in pain. Compared to other ways of measuring pain-related thoughts, this questionnaire is unique in that the individual does not need to be in pain while completing it.
Anxiety and Depression | Baseline
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No